CLINICAL TRIAL: NCT05108077
Title: Treatment of Metastatic Tumors of the Urogenital Area (Bladder Cancer, Renal Cancel) With Cytokine-induced Killer Cells
Brief Title: Treatment of Metastatic Tumors of the Urogenital Area With Cytokine-induced Killer Cells
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus (Other Government)
Collaborators: Belarusian State Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBCE_CIK
Record Dates: First submitted 2021-09-22; First posted 2021-11-04 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Bladder Cancer; Renal Cancer
Keywords: Bladder Cancer; Renal Cancer; CIK
MeSH Terms: conditions — Urinary Bladder Neoplasms; Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cytokine-induced killer cells (Experimental): Patients with the metastatic tumors of the urogenital area receiving standard treatment and autologous cytokine-induced killer cells
  Interventions: Biological: cytokine-induced killer cells; Other: Standard treatment according to the Clinical protocols
- Control (Active Comparator): Patients with metastatic tumors of the urogenital area receiving standard treatment
  Interventions: Other: Standard treatment according to the Clinical protocols

INTERVENTIONS:
Biological: cytokine-induced killer cells — Autologous cytokine-induced killer cells injected intravenously
  Arms: Cytokine-induced killer cells
Other: Standard treatment according to the Clinical protocols — Standard treatment of bladder/renal cancer according to the Clinical protocols

SUMMARY:
Treatment of metastatic tumors of the urogenital area with cytokine-induced killer cells

DETAILED DESCRIPTION:
Treatment of metastatic tumors of the urogenital area using autologous cytokine-induced killer cells

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of pTa metastatic tumors of the urogenital area;
* Patient who require repetitive transurethral resection;
* Expression of muc-1/wt-1 by the tumor;
* EGOC 0-3;

Exclusion Criteria:

* any medical condition which can be associated with the high risk for the patient;
* pregnancy/lactation;
* chronic infections, including hepatitis B/C, tuberculosis, HIV

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The relapse-free survival | 1 year
  The duration of relapse-free survival
The relapse-free survival | 2 year
  The duration of relapse-free survival
The relapse-free survival | 3 year
  The duration of relapse-free survival
Adverse effects associated with the therapy | 1 month
  Determination of adverse effects associated with the therapy
Adverse effects associated with the therapy | 1 year
  Determination of adverse effects associated with the therapy

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Hancharou, Study Director — the Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus; Alexander Prokhorov, Dr, Study Director — Belarusian State Medical University
Locations (1):
- Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus, Minsk, Belarus

IPD SHARING:
Plan to Share IPD: No